CLINICAL TRIAL: NCT04392778
Title: What is the Effect of Mesenchymal Stem Cell Therapy on Seriously Ill Patients With Covid 19 in Intensive Care? (Prospective Double Controlled Study)
Brief Title: Clinical Use of Stem Cells for the Treatment of Covid-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SBÜ Dr. Sadi Konuk Eğitim ve Araştırma Hastanesi (Other)
Collaborators: Istinye University (Other); Regenerative Medicine and Stem Cell Production Center Liv MedCell (Unknown); Liv Hospital (Ulus) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bak. Sadi Konuk-Istinye Uni.
Record Dates: First submitted 2020-04-25; First posted 2020-05-19 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2020-05

CONDITIONS: Covid19; Pneumonia; Multiple Organ Failure; Corona Virus Infection
Keywords: Covid-19; Pneumonia; Multiple Organ Failure; Coronavirus; Mesenchymal stem cells; Cellular therapy
MeSH Terms: conditions — COVID-19; Pneumonia; Multiple Organ Failure; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Untreated (No Intervention): Group 1: patients that are not on a ventilator (n=10) No extra intervention will be done.
- Saline Control (Sham Comparator): Group 2: patients that are on a ventilator and will receive saline injections (n=10) as control for MSC transplantation group (3).
  Interventions: Biological: Saline Control
- Experimental UC-MSCs (Experimental): Group 3: patients that are on a ventilator and will receive MSC transplantation injections (n=10)
  Interventions: Biological: MSC Treatment

INTERVENTIONS:
Biological: MSC Treatment — Protocol length: 1 week
  Doses:
  1. Application: 3 million cells/kg IV-------------------------------------------------0 day
  2. Application: 3 million cells/kg IV ------------------------------------------------3rd day
  3. Application: 3 million cells/kg IV -------------------------------------------------6th day
  will be given to patients positively, clinically and radiologically diagnosed with COVID-19, followed with 3 months observation.
  Arms: Experimental UC-MSCs
Biological: Saline Control — Saline will be given to patients positively, clinically and radiologically diagnosed with COVID-19, followed with 3 months observation.
  Arms: Saline Control

SUMMARY:
This study aims to use the regenerative and repair abilities of stem cells to fight against the harmful effects of the novel coronavirus Covid-19 and therefore develop a treatment strategy. It is known that fatalities from this virus is largely caused by its damage to lungs and other organs. As the disease progresses, these organs fail and lead to mortality. Our hope is that the stem cell transplantation from healthy donors will repair the damage caused by the virus and result in a healthy recovery.

DETAILED DESCRIPTION:
Introduction:

The COVID-19 corona virus epidemic has spread from Wuhan, China to the whole world, and has been declared a pandemic by WHO worldwide. In severe patients, ARDS and multiple organ failure can be seen. This condition is associated with cytokine storm in the body. When the virus invades the body, dentric cells can activate macrophages, lymphocytes and natural killer cells. Mesenchymal stem cells (MKH) not only inhibit the abnormal activation of T lymphocytes and macrophages, but also encourage them to differentiate into regulatory T cell subsets (Treg) clusters and anti-inflammatory macrophages. MSCs application proved therapeutic efficiency during influenza infection resulting in reduced impairment of alveolar fluid clearance and lung injury. This was attributed towards attenuation of pro-inflammatory cytokine secretion, inflammatory cell recruitment and increased alveolar macrophages content.

Aim of study:

1. To provide immune modulation to patients with COVID-19 who are taken to intensive care and resistant to treatment by performing MSCs transplantation and to reduce the damage caused by cytokin storm to tissues and organs,
2. Correcting immunosuppression in patients and increasing the fight against COVID-19 virus by CD4+T, CD+8T cellular cell arrangement,
3. It is to accelerate the recovery in organ damage by increasing growth factors by means of MSCs.

Materials and method:

Patients diagnosed with COVID-19 infection as clinically, radiologically and laboratory-wise will be divided into three groups:

Group 1: patients that are not on a ventilator (n=10) Group 2: patients that are on a ventilator and will receive saline injections (n=10) Group 3: patients that are on a ventilator and will receive MSC transplantation injections (n=10)

Mesenchymal stem cells originating from allogenic umbilical cord produced under GMP conditions will be administered in 3 times, with doses indicated below, intravenously within 1 week.

Dose:

1. Application: 3 million cells / kg IV ---------------------------------------- --------- 1 day
2. Application: 3 million cells / kg IV ---------------------------------------- --------- 3. Day
3. Application: 3 million cells / kg IV ---------------------------------------- --------- 6. Day

The blood will be analyzed for the expression levels of growth factors, including vascular endothelial growth factor, fibroblast growth factor, platelet derived-growth factor, epidermal growth factor, transforming growth factor beta, hepatocyte growth factor, nerve growth factor, VEGF receptor (VEGFR), angiopoietin1 (Angpt-1), and Angpt-2, using sandwich enzyme-linked immune sorbent assays (ELISAs). Investigators also analyzed the caspase-3 system in the blood. immunoassay kits will be used for analyses in accordance with the manufacturer's instructions.

Biochemical parameters of the liver, such as alanine transaminase (ALT), aspartate transaminase (AST), total protein, albumin, total bilirubin, direct bilirubin, and alkaline phosphatase (ALP) levels, will be measured in the venous blood samples.

Proinflammatory (IL1-β, IL-6, TNFα, INF-γ) and anti-inflammatory (IL-2, IL-4, IL-10, IL-13) cytokines will be examined in venous blood in order to determine the immune modulatory effect of stem cells. CD4 + T, CD4 + T killer cells Granulocyte macrophage colony factor BLC-2 VEGF-R angiopoetin-1, angiopoetin-2 Total antioxidant capacity (TAC) Total oxidant capacity (TOC).

ELIGIBILITY:
Inclusion Criteria:

* 40-60 years old male or female
* Confirmed 2019-nCoV infection with RT-PCR Laboratory test
* Confirmed Pneumonia with chest radiography and computer tomography
* and any of the following criteria:

  1. Shortness of breath (RR ≥30/min)
  2. Resting finger oxygen saturation 93%
  3. Arterial oxygen partial pressure (PaO2)/oxygen absorption concentration (FiO2) ≤ 300MMHG
  4. Advancing of focus in Pulmonary imaging to >50% in 24-48 hours

Exclusion Criteria:

* Those who are not pregnant, breastfeeding and pregnant but who do not take effective contraceptive measures;
* Patients with malignant tumors, other serious systemic diseases and psychosis;
* Informed consent is not given or does not comply with the test requirements.
* Co-infection of HIV, tuberculosis, influenza virus, adenovirus and other respiratory infection virus.
* Pneumonia caused by bacteria, mycoplasma, chlamydia, legionella, fungi or co-infection of HIV, tuberculosis, influenza virus, adenovirus and other respiratory infection virus.
* Obstructive HABP / VABP caused by lung cancer or other known causes; Long-term history of use of immunosuppressive agents;
* History of epilepsy and need for continuous anticonvulsant therapy or anticonvulsant therapy taken within 3 years;
* Invasive ventilation
* Shock
* Other organ failures

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | 3 months
  Improvement of clinical symptoms related to Covid-19 infection (fever, pneumonia, shortness of breath)

SECONDARY OUTCOMES:
Lung damage improvement | 3 months
  Improvement of lungs assessed by CT Scan
Sars-Cov-2 viral infection laboratory test | 3 months
  Negative, measured by RT-PCR laboratory tests for the virus
Blood test | 3 months
  Cell types and numbers

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan T Adas, Prof.Dr., Principal Investigator — SBÜ Dr. Sadi Konuk Eğitim ve Araştırma Hastanesi; Erdal Karaoz, Prof.Dr., Principal Investigator — Istinye University
Locations (2):
- Turkey (Türkiye) (2):
  - Istinye University, Istanbul
  - SBÜ Dr. Sadi Konuk Eğitim ve Araştırma Hastanesi, Istanbul

IPD SHARING:
Plan to Share IPD: No